CLINICAL TRIAL: NCT04448002
Title: AIM2ACT: A Mobile Health Tool to Help Adolescents Self-Manage Asthma
Acronym: AIM2ACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202000748; R01HL153119 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: Adolescent
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Block randomization will ensure a 1:1 ratio
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIM2ACT (Experimental): AIM2ACT is the experimental arm for the trial. AIM2ACT is a dyadic mHealth intervention designed to sustain caregiver involvement and monitoring as well as guide dyads through collaborative asthma management.
  Interventions: Behavioral: AIM2ACT
- mHealth Attention Control Condition (Active Comparator): The mHealth attention control condition is the active comparator arm in the trial that accounts for staff attention and novelty of technology based asthma management intervention.
  Interventions: Behavioral: mHealth Attention Control Condition

INTERVENTIONS:
Behavioral: AIM2ACT — AIM2ACT is a mobile health tool that is designed to facilitate collaborative asthma management between early adolescents and their caregivers. AIM2ACT contains the following components: 1) ecological momentary assessment to identify personalized strengths and weaknesses in asthma self-management behaviors; 2) collaborative identification and tracking of goals that help early adolescents to become increasingly independent in managing their asthma; and 3) a suite of engaging skills training videos to help dyads understand how to use AIM2ACT and work together to set asthma self-management goals, develop and achieve the goals articulated in a behavioral contract, and engage in problem-solving communication.
  Arms: AIM2ACT
Behavioral: mHealth Attention Control Condition — Dyads in the mHealth attention control condition will not receive personalized asthma management feedback, will not be guided through collaborative identification and tracking of asthma self-management goals, and will not have access to skills training videos. Instead, dyads will receive static educational information on their smartphones about behavioral management techniques they can use to target improving asthma self-management.
  Arms: mHealth Attention Control Condition

SUMMARY:
The aim is to test the efficacy of AIM2ACT and long-term maintenance of treatment effects in a fully-powered randomized controlled trial with 160 early adolescents with poorly controlled persistent asthma, ages 12-15 years, and a caregiver

ELIGIBILITY:
Inclusion criteria are:

1. Adolescent is 12-15 years old
2. Caregiver is between 18-70 years-old
3. Adolescent lives in the residence of caregiver
4. Adolescent and caregiver can speak and read English
5. (a) Adolescent has been diagnosed as having asthma, OR (b) Doctor has stated the adolescent has asthma, OR (c) Adolescent has had breathing problems in the past 12 months
6. Adolescent has had an active inhaled corticosteroid prescription for ≥ 4 weeks
7. (a) During the past 14 days (that is, during the past fourteen 24-hour periods that include daytime and nighttime), the adolescent has experienced one or more of the following: (i) Asthma symptoms such as wheezing, shortness of breath, or tightness in the chest, or cough on more than 4 separate days; (ii) Woken up because of asthma symptoms such as wheezing, shortness of breath, or tightness in the chest, or cough on 1 or more separate nights; (iii) Had to slow down or stop play or usual activities or missed school because of asthma, wheezing, or tightness in the chest, or cough on more than 4 separate days; (iv) Used any asthma rescue medicine (sometimes called a quick relief medicine) on more than 4 separate days

   * OR

     (b) In the past year, adolescent has had one or more of the following: (i) 2 or more exacerbations requiring oral systemic corticosteroids; (ii) 2 or more emergency department visits; (iii) 1 hospitalization; (iv) 2 or more urgent medical care visits due to asthma
   * OR

     (c) Adolescent scores 19 or lower on the Asthma Control Test

Exclusion criteria are -

Families will be excluded if:

1. The family is currently involved in an asthma management intervention above and beyond usual care, OR
2. Adolescent is unable to complete study procedures independently.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control using asthma control questionnaire | Change in baseline, post-intervention,3 months, and 6 months, and 12 month follow-up
  Measured via the Asthma Control Test questionnaire which has 5 items that assesses frequency of daytime and nocturnal asthma symptoms, activity limitations, and perceptions of disease control.Adolescents will complete all 5 items independently of caregivers. Scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma."

CONTACTS AND LOCATIONS:
Overall Officials: Sreekala Prabhakaran, M.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health Pediatrics, Gainesville, Florida
  - Nemours Children's Hospital, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fedele DA, Thomas JG, McQuaid EL, Gurka M, Berg CA, Prabhakaran S. AIM2ACT: Randomized controlled trial protocol for a mobile health intervention for early adolescents with asthma. Contemp Clin Trials. 2022 Dec;123:107011. doi: 10.1016/j.cct.2022.107011. Epub 2022 Nov 15. PMID 36396068